CLINICAL TRIAL: NCT00880724
Title: European Post Market Study: A Prospective, Randomized, Controlled, Multicenter Study to Evaluate the Performance of the IBV Valve System for the Treatment of Severe Emphysema
Brief Title: European Multi-center Post Market Study of the IBV Valve System
Acronym: IBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-01576 AD
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2009-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Emphysema; Bronchoscopic Treatment; Interventional Bronchoscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medical management (No Intervention)
  Interventions: Device: IBV Valve

INTERVENTIONS:
Device: IBV Valve — Placement of IBV Valve in the airways of treatment subjects. Bronchoscopic procedure in control group.
  Other Names: BLVR; Endoscopic Volume Reduction; Endobronchial Valve

SUMMARY:
The objective of this randomized, blinded, multicenter, controlled study is to compare the performance of the IBV Valve System (treatment group) to a control group receiving a sham bronchoscopy procedure without valve placement.

DETAILED DESCRIPTION:
The IBV Valve System (Spiration Inc. Redmond, WA) has CE Mark approval for the treatment of diseased and damaged lung. The devices are one-way valves that can be placed in the airways via flexible bronchoscopy limiting airflow distally. For the treatment of emphysema, valves are placed in airways communicating to the most diseased areas of lung tissue to re-direct airflow to less diseased areas. A multicenter, blinded and randomized study of these valves is being conducted in 7 centers in 6 European countries. The study is evaluating the effectiveness of this therapy for the treatment of upper lobe predominant emphysema in patients with severe to very severe emphysema (GOLD classification 3 to 4) that despite best medical management continue having poor quality of life, severe symptoms and physical limitations. The primary endpoints are to measure and compare responses using the St. George's Respiratory Questionnaire and lung volume changes as measured by CT-scans. Consented patients that meet the strict inclusion criteria have a bronchoscopic procedure and are randomized into treatment or control (no valves) groups. After the procedure, all patients stay blinded to their group assignment and have follow-up evaluations at 1 and 3 months. After the 3-month evaluation, each patient is un-blinded. The treatment group is then scheduled for an additional follow-up at 6 months and the control group is offered valve treatment (rollover) and evaluated approximately 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 74 years of age
* Predominantly upper lobe emphysema and severe dyspnea
* Satisfies the criteria of the ATS/ERS Guidelines for Management of Stable COPD
* Physical ability to participate in the study by performing a 6-minute walk distance of > 140m
* No cigarette smoking for 4 months and willing to abstain throughout the study
* Severe airflow obstruction defined by FEV1 45% of predicted
* Severe hyperinflation defined by: TLC > 100% of predicted and RV > 150% of predicted

Exclusion Criteria:

* Between 70 and 74 years of age and an FEV1 or DLCO < 20% of predicted
* Severe gas exchange abnormalities
* Major medical disease that will limit evaluation, participation or follow-up
* Active asthma component to their disease
* Giant bulla (> 1/3 volume of lung)
* Severe pulmonary hypertension
* Requirement for > 6L02 to keep saturation > 90% with exercise
* Evidence of systemic disease or neoplasia expected to compromise survival during the 6-month study period

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The difference between the response rates of the treatment and control groups. | 3-months post randomization

CONTACTS AND LOCATIONS:
Locations (7):
- Landeskrankenhaus, Innsbruck, Austria
- CHU Saint Pierre, Brussels, Belgium
- Medizinische Hochschule Hannover, Hanover, Germany
- Spedali Civili di Brescia, Brescia, Italy
- Spain (2):
  - Bellvitge Hospital, Barcelona
  - Clinica Universitaria de Navarra, Pamplona
- Royal Preston Hospital/Lancashire Teaching Hospitals, Preston, United Kingdom

REFERENCES:
- [Derived] Ninane V, Geltner C, Bezzi M, Foccoli P, Gottlieb J, Welte T, Seijo L, Zulueta JJ, Munavvar M, Rosell A, Lopez M, Jones PW, Coxson HO, Springmeyer SC, Gonzalez X. Multicentre European study for the treatment of advanced emphysema with bronchial valves. Eur Respir J. 2012 Jun;39(6):1319-25. doi: 10.1183/09031936.00019711. PMID 22654006
- See also: Sponsor website — http://www.spiration.com